CLINICAL TRIAL: NCT01548807
Title: Phase 1 Trial of the Mammalian Target of Rapamycin (mTOR) Inhibitor Everolimus Plus Radiation Therapy (RT) for Salvage Treatment of Biochemical Recurrence in Prostate Cancer Patients Following Prostatectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: UPCC 06810
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer Patients With Detectable PSA Following Prostatectomy
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Everolimus (RAD001)

SUMMARY:
This is a Phase 1 dose escalation study of an investigational agent, everolimus, given in combination with standard radiation therapy, in prostate cancers with a rising PSA following a prostatectomy. A maximum of 33 people will be enrolled on this study at the University of Pennsylvania. The primary objective of this study is to determine the acute and chronic toxicities and maximum tolerated dose of everolimus with concurrent radiation.

ELIGIBILITY:
Inclusion Criteria:

* - Patient must have a history of prostatectomy (Open Radical or Robotic Assisted) with histopathologic documentation of adenocarcinoma of the prostate
* Patient must have biochemical evidence of PSA including one of the following: a). biochemical recurrence (defined as nadir + 2 rises measured at least 2 weeks apart) and b). PSA doubling time of less than or equal to 6 months; OR c). persistently elevated PSA(PSA post prostatectomy of 0.2 ng/mL if standard assay or greater than 0.05 if ultrasensitive PSA assay)
* Patient must be a candidate for salvage radiotherapy to the prostate bed
* Age greater or equal to 18 years
* ECOG performance status less than or equal to 1
* Adequate bone marrow function
* Adequate liver and renal function Adequate renal function: serum creatinine 1.5 x ULN
* Signed informed consent
* Patient must have archival prostate tumor block available for analysis of correlatives

Exclusion Criteria:

* - Indication for lymph node radiation (i.e. evidence of LB node metastases)
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 4 weeks
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated liver vaccines within one week of study entry or during study period. Close contact with those who have received attenuated liver vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  1. . Symptomatic congestive heart failure of New York heart Association Class III or IV
  2. . unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  3. . severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
  4. . uncontrolled diabetes
  5. . active (acute or chronic) or uncontrolled severe infections
  6. . liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).

Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.

* A known history of HIV seropositivity as everolimus has immunosuppressant properties
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to everolimus (RAD001) or other rapamycins (sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Male patient whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-09; Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Number of Participannts with Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Haas, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States